CLINICAL TRIAL: NCT05838105
Title: Prospective Randomized Control Study of Two Different Types of Luteal Phase Support in Natural Cycle Frozen Embryo Transfer and Its Effect on Pregnancy Rates
Brief Title: Two Different Types of Luteal Phase Support in Natural Cycle Frozen Embryo Transfer and Its Effect on Pregnancy Rates
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Heli Alexandroni, Alexandroni Heli, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LutealSupport
Record Dates: First submitted 2023-04-20; First posted 2023-05-01 (Actual); Last update posted 2023-05-01 (Actual); Status verified 2023-04

CONDITIONS: Luteal Phase Support
MeSH Terms: interventions — Gonadotropin-Releasing Hormone; Progesterone

STUDY DESIGN:
Intervention Model Description: All patients will be randomly divided into two groups, each will receive a different luteal treatment:
  1. Study group - patients will receive luteal support with GNRH agonist and HCG according to departmental protocol (described later).
  2. Control group - patients will receive luteal support with vaginal progesterone.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Active Comparator): Patients will receive luteal support with GNRH agonist and HCG according to departmental protocol:
  Cleavage stage embryo:
  * ET day (embryo day 2-3) - Ovitrelle 125mcg
  * Day 3 after ET - Ovitrelle 125mcg + Decapeptyl 0.1mg
  * Day 6 after ET- Ovitrelle 125mcg
  * Day 9 after ET - Ovitrelle 125mcg
  Embryo blastocyst stage:
  * ET day (embryo day 5-6) - Ovitrelle 125mcg + Decapeptyl 0.1mg
  * Day 3 after ET - Ovitrelle 125mcg
  * Day 6 after ET - Ovitrelle 125mcg
  Interventions: Drug: GnRH agonist; Drug: hCG
- Control group (Active Comparator): Patients will receive luteal support with vaginal progesterone - 100 mg Endometrin twice daily until week 8 of pregnancy.
  Interventions: Drug: Progesterone 100Mg Vag Tab

INTERVENTIONS:
Drug: GnRH agonist — 125 mcg once at the day mentioned
  Arms: Study group
Drug: hCG — dose as mentioned
  Arms: Study group
Drug: Progesterone 100Mg Vag Tab — dose as mentioned
  Arms: Control group

SUMMARY:
The aim of the study is to compare the pregnancy rate between women treated with Gonadotropin Releasing Hormone (GnRH) agonist together with Human Chorionic Gonadotropin (HCG) and standard luteal support with progesterone following transfer of frozen embryos in in-vitro-fertilization (IVF) natural cycles.

DETAILED DESCRIPTION:
The rate of frozen embryos transfer (FET) has increased in recent years due to a higher tendency of single embryo transfer, use of preimplantation genetic testing, and prevention of ovarian hyperstimulation.

There are different methods to prepare the endometrium for FET:

1. Natural cycle (NC) - natural preparation of the body for implantation without the need for medicinal intervention.
2. Modified natural cycle (mNC) - Inducing ovulation by administration of Human Chorionic Gonadotropin (HCG) trigger.
3. Medical - preparation of endometrium with hormones (estrogen and progesterone).

Following embryo transfer, luteal phase support should be considered. Administration of treatment depends on the type of cycle chosen (either natural or medicated). Treatment options include progesterone, HCG and Gonadotropin Releasing Hormone (GnRH) analog - either one of them or combined. Different protocols (dosages and duration of use) with different pregnancy outcomes were explore before with inconclusive results. We wish to investigate administration of GnRH agonist+HCG vs. progesterone.

Patients included in the study will be women undergoing natural cycle FET at the IVF center in Shaare Zedek, Jerusalem, Israel. All patients will be randomly divided into two groups, each will receive a different luteal treatment support as will be detailed later. Patients demographic data and pregnancy outcomes will be collected.

Based on the clinical pregnancy rate in the prospective study by Bjuresten, et al [Fertil Steril, 2011], where a clinical pregnancy rate of 32% was found among women treated with progesterone for luteal support, and given an alpha of 5% and a power of 80%, 144 women (72 women in each group) are required in order to demonstrate a clinical pregnancy rate of 55% in the study group.

Comparison of categorical variables will be carried out using the the chi-squared test. Comparison of continuous variables will be performed using the Students t-Test or Mann-Whitney U method depending on the variable distribution (normal vs. non-normal distribution, respectively). A multivariate regression will also be conducted in order to determine which variables are significantly and independently related. Statistical significance will be defined when P values are less than 0.05

ELIGIBILITY:
Inclusion Criteria:

* Normo-ovulatory women
* Women undergoing frozen embryos transfer in a natural cycle
* Age 18-45
* BMI 18-35

Exclusion Criteria:

* Women undergoing medicated frozen embryos transfer
* Women with a BMI over 35 or under 18.
* Women with hydrosalpinges
* Women with defects or uterine malformations (congenital) or acquired such as myomas
* Egg donation and surrogacy
* Use of preimplantation genetic testing

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — patients going in-vitro-fertility treatments with embryo transfer
Enrollment: 144 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | up to two month after embryo transfer
  visualization of intrauterine gestational sac on ultrasound divided by number of transfers

SECONDARY OUTCOMES:
Overall pregnancy rate | up to two month after embryo transfer
  number positive beta-hCG divided by total number of transfers
Implantation rate | up to two month after embryo transfer
  number of gestational sacs divided by number of embryos transferred
Ectopic pregnancy rate | up to two month after embryo transfer
  number of ectopic pregnancy divided by number of positive beta-hCG
Miscarriage rate | up to 20 weeks after embryo transfer
  number of non-viable before 24 weeks divided by total number of positive beta-hCG
Live birth rate | up to 42 weeks after embryo transfer
  number of live births after 24 weeks divided by number of transfers.

CONTACTS AND LOCATIONS:
Overall Officials: Keren Rotshenker Olshnika, MD, Principal Investigator — Sharee Zedek Medical Center, Israel
Locations (1):
- Shaare Zedek medical center, Jerusalem, Israel

REFERENCES:
- [Background] Groenewoud ER, Cantineau AE, Kollen BJ, Macklon NS, Cohlen BJ. What is the optimal means of preparing the endometrium in frozen-thawed embryo transfer cycles? A systematic review and meta-analysis. Hum Reprod Update. 2013 Sep-Oct;19(5):458-70. doi: 10.1093/humupd/dmt030. Epub 2013 Jul 2. PMID 23820515
- [Background] Le Lannou D, Griveau JF, Laurent MC, Gueho A, Veron E, Morcel K. Contribution of embryo cryopreservation to elective single embryo transfer in IVF-ICSI. Reprod Biomed Online. 2006 Sep;13(3):368-75. doi: 10.1016/s1472-6483(10)61441-1. PMID 16984767
- [Background] Loutradi KE, Kolibianakis EM, Venetis CA, Papanikolaou EG, Pados G, Bontis I, Tarlatzis BC. Cryopreservation of human embryos by vitrification or slow freezing: a systematic review and meta-analysis. Fertil Steril. 2008 Jul;90(1):186-93. doi: 10.1016/j.fertnstert.2007.06.010. Epub 2007 Nov 5. PMID 17980870
- [Background] Weissman A, Horowitz E, Ravhon A, Steinfeld Z, Mutzafi R, Golan A, Levran D. Spontaneous ovulation versus HCG triggering for timing natural-cycle frozen-thawed embryo transfer: a randomized study. Reprod Biomed Online. 2011 Oct;23(4):484-9. doi: 10.1016/j.rbmo.2011.06.004. Epub 2011 Jun 15. PMID 21840758
- [Background] Mackens S, Stubbe A, Santos-Ribeiro S, Van Landuyt L, Racca A, Roelens C, Camus M, De Vos M, van de Vijver A, Tournaye H, Blockeel C. To trigger or not to trigger ovulation in a natural cycle for frozen embryo transfer: a randomized controlled trial. Hum Reprod. 2020 May 1;35(5):1073-1081. doi: 10.1093/humrep/deaa026. PMID 32395750
- [Background] Ghobara T, Gelbaya TA, Ayeleke RO. Cycle regimens for frozen-thawed embryo transfer. Cochrane Database Syst Rev. 2017 Jul 5;7(7):CD003414. doi: 10.1002/14651858.CD003414.pub3. PMID 28675921
- [Background] Montagut M, Santos-Ribeiro S, De Vos M, Polyzos NP, Drakopoulos P, Mackens S, van de Vijver A, van Landuyt L, Verheyen G, Tournaye H, Blockeel C. Frozen-thawed embryo transfers in natural cycles with spontaneous or induced ovulation: the search for the best protocol continues. Hum Reprod. 2016 Dec;31(12):2803-2810. doi: 10.1093/humrep/dew263. Epub 2016 Oct 25. PMID 27798046
- [Background] Fatemi HM, Kyrou D, Bourgain C, Van den Abbeel E, Griesinger G, Devroey P. Cryopreserved-thawed human embryo transfer: spontaneous natural cycle is superior to human chorionic gonadotropin-induced natural cycle. Fertil Steril. 2010 Nov;94(6):2054-8. doi: 10.1016/j.fertnstert.2009.11.036. Epub 2010 Jan 25. PMID 20097333

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/05/NCT05838105/Prot_SAP_000.pdf